CLINICAL TRIAL: NCT04862195
Title: Double-blinded, Randomized, Adaptive Registrational Trial to Compare Effectiveness of Two Digital Software Medical Devices (Attune™ and Cerena™) as Interventions for Physical and Emotional Health in Adjunctive Oncology Treatment
Brief Title: Registrational Trial to Compare Effectiveness of Two Digital Software Medical Devices as Adjunctive Oncology Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was halted prematurely due to slow enrollment
Sponsor: Blue Note Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROT001
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attune™ (Active Comparator): Attune™ is a completely digital, 10-session, cognitive behavioral therapeutic intervention.
  Interventions: Device: Attune™
- Cerena™ (Active Comparator): Cerena™ is a completely digital, 10-session, health education and wellness intervention.
  Interventions: Device: Cerena™

INTERVENTIONS:
Device: Attune™ — Software as a medical device
  Arms: Attune™
Device: Cerena™ — Software as a medical device
  Arms: Cerena™

SUMMARY:
This is a non-significant risk, double-blinded, randomized, registrational study to compare the effectiveness of two digital, software only, medical devices (SaMD) (attune™ and cerena™) in reducing cancer-related anxiety and depression symptoms when used adjunctively with multidisciplinary (medical, psychosocial) oncology usual care regimens for up to 10 weeks.

Study population will consist of up to 553 participants with stage I-III breast cancer or stage I-III NSCLC. The primary endpoint is percent improvement in anxiety symptoms at Week 10 and secondary endpoints of percent improvement in depressive symptoms will be assessed at Week 12.

An interim analysis for efficacy and futility will be conducted once 236 participants have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer or Stage I-III NSCLC who are currently in active treatment or have completed initial cancer directed treatments (surgery, radiation, chemotherapy) within the past 3 months;
* Are experiencing at least moderate anxiety (GAD-7 >10) or mild-to-moderate depression (PHQ-8 score 5-11);
* Are fluent in English; and
* Have access to smartphone, or tablet capable of running iOS or Android software.

Exclusion Criteria:

* Previous history of cancer;
* <2-yr survival prognosis as determined by treating clinician;
* Currently participating in investigative CBT trial for treatment of anxiety or depression;
* Participant is unable to complete training, has cognitive deficits, more severe psychiatric conditions, lack of access to internet accessible device or psycho-social conditions (e.g., other social conditions, that would interfere with adherence to self-directed care), such that in investigator's opinion the participant would be unable to complete the study;
* Recently completed use of Blue Note Therapeutics Covid Cancer Care Program or other Blue Note Therapeutics-sponsored study; and
* PHQ-9 Q9 response >0 AND Columbia Suicide Severity Risk Scale (or equivalent) score of Category 2- "suicidal ideation" at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Cancer-related symptoms of anxiety (1) | Baseline up to Week 10
  Percent reduction in PROMIS-A scores, reduction indicates reduced anxiety

SECONDARY OUTCOMES:
Cancer-related symptoms of depression (1) | Baseline up to Week 10
  Percent reduction in PROMIS-D scores, reduction indicates reduced depression
Cancer-related symptoms of anxiety (2) | Baseline up to Week 12
  Percent reduction in PROMIS-A scores, reduction indicates reduced anxiety
Cancer-related symptoms of anxiety (3) | Baseline up to Week 10
  Percent reduction in Clinical Global Impression Scale and Improvement scores, reduction indicates reduced anxiety
Cancer-related symptoms of depression (4) | Baseline up to Week 12
  Percent reduction in Clinical Global Impression Scale and Improvement scores, reduction indicates reduced depression
Mean mHealth App Usability Questionnaire (MAUQ) for Standalone mHealth Apps Used by Patients | Baseline up to Week 10
  Higher scores indicate higher ease of use / easier to use applications

OTHER OUTCOMES:
Quality of life via PROMIS-Global Health v1.2 | Weeks 10 and Week 12
  The PROMIS Global Health measures assess an individual's physical, mental, and social health. The measures are generic, rather than disease-specific, and often use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health (Promis-Global Health Scoring Manual, 2017). Higher scores for responses always indicate better health.
Patient self-efficacy via the Patient Activation Measure-13 (PAM-13) | Weeks 10
  Patient Activation Measures-the knowledge, skills, and confidence to manage one's health is associated with improved self-management behaviors in cancer patients. A patient activation measure (PAM) using PAM-13 will be used to assess participant engagement at baseline after PROMIS-A and PROMIS-D are completed and at Week 10. Higher scores indicate higher self-efficacy.
Patient self-efficacy via the Measurement of Current Status (MOCS) Part A and Part B | Baseline, Week 6, and Week 10
  The Measure of Current Status (MOCS) scale comes from research on the effects of a multi-modal cognitive-behavioral stress management intervention on the psychosocial well-being of cancer patients. The MOCS has two sections. Part A is items measuring participants' current self-perceived status on several skills that are targeted by the intervention: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Part B assesses potential "nonspecific effects" of the intervention: feelings of normalcy vs. alienation, sense of cohesiveness with other patients, perceptions of care from persons around them, and a sense of being better off than other cancer patients. All items were framed in such a way that they are sensible to participants in both conditions. MOCS measurements will be taken at Baseline, Week 6, and Week 10. Higher scores indicate higher self-efficacy.
Immune cell transcription | Baseline up to Week 12
  Analyses will focus on inflammatory gene expression and related gene regulation pathways due to their established relevance for disease progression/recurrence in the aftermath of cancer diagnosis and treatment, and their role in promoting symptoms of depression or anxiety via effects on central nervous system function

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Ganz, MD, Principal Investigator — University of California, Los Angeles
Locations (13):
- United States (13):
  - OPN Healthcare, Glendale, California
  - Oncology Physicians Network Healthcare, Los Alamitos, California
  - Redlands Oncology, Redlands, California
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Illinios Cancer Care, Peoria, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rogel Cancer Center | University of Michigan, Ann Arbor, Michigan
  - SCL Health, Billings, Montana
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - New York Cancer & Blood Specialists, Port Jefferson Station, New York
  - Tri-County Hematology and Oncology-Massillon, Massillon, Ohio
  - MD Anderson, Houston, Texas
  - Northwest Medical Specialty, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No